CLINICAL TRIAL: NCT03312959
Title: Heavy Bupivacaine Versus Plain Bupivacaine in Peribulbar Block
Brief Title: Heavy Bupivacaine in Peribulbar Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: badway 2
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Anesthetics, Local
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperbaric bupvacaine group (Experimental): Peribulbar block will be performed using a total volume of 7 ml 6ml hyperbaric bupivacaine 0.5% + hyaluronidase (50 IU) in 1ml saline
  Interventions: Drug: hyperbaric bupvacaine in Peribulbar block
- isobaric bupvacaine group (Active Comparator): Peribulbar block will be performed using a total volume of 7 ml 6ml isorbaric bupivacaine 0.5% + hyaluronidase (50 IU) in 1ml saline
  Interventions: Drug: isobaric bupvacaine in Peribulbar block

INTERVENTIONS:
Drug: hyperbaric bupvacaine in Peribulbar block — hyperbaric bupivacaine in Peribulbar block will be injected in the posterior segment surgery
  Other Names: trial group
  Arms: hyperbaric bupvacaine group
Drug: isobaric bupvacaine in Peribulbar block — isobaric bupivacaine in Peribulbar block will be injected in the posterior segment surgery
  Other Names: control group
  Arms: isobaric bupvacaine group

SUMMARY:
Most of the ophthalmic procedures are performed under local anesthesia as the patient is often elderly and with diseases. This may increase the risk of morbidity and mortality under general anesthesia. Different eye blocks have been practiced with great success. Moreover, it is associated with less hemodynamic instability, less respiratory depression, better postoperative pain relief, and less nausea and vomiting than general anesthesia. It is also associated with a reduction in stress response, maintained oxygen saturation and cardiovascular stability, in addition to the production of good akinesia and anesthesia alleviating occulo-medullary reflexes, all make local anesthesia more superior and safe technique.

DETAILED DESCRIPTION:
Peribulbar anesthesia is widely practiced now as a safe local block for cataract eye surgeries. However, the limited duration of these blocks was shown to be the main problem encountered intra-operatively. Therefore, additional top-up doses are usually needed to continue the operation. Many kinds of research tried to introduce solutions in order to prolong the duration of the local anesthetics used. Many researchers tried different volumes, doses and adjuvant to local anesthetics, and studied their effects There are many studies that evaluated the effect of baricity of local anesthetic on the potency of motor block and the duration of motor and sensory blockade.

However, no properly designed randomized, controlled studies have evaluated the feasibility and reliability of baricity local anesthetic agents used for the peribulbar block.

Aim of the work prospective, randomized study was conducted to evaluate the effects of the baricitized bupivacaine used for the peribulbar block in patients undergoing posterior segment surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiology (ASA) I or II.
* 30-80 years old
* Patients scheduled for elective unilateral posterior segment surgeries.

Exclusion Criteria:

* Patient's refusal.
* orbital deformity
* axial length( >28 mm )
* increased intraocular pressure, or if they were blind in the contralateral eye, international normalized ratio (INR) > 1.5
* allergy to local anesthetics, mentally retarded patients

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-01-20 (Estimated); Study Completion 2018-01-31 (Estimated)

PRIMARY OUTCOMES:
The onset and duration of lid and globe akinesia | 12 hours postoperative
  scoring the ocular movements in each direction of gaze

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No